CLINICAL TRIAL: NCT03348813
Title: HIV/STI Prevention Among Black Adolescents With Mental Illnesses
Brief Title: HIV/STI Prevention Among Black Adolescents With Mental Illnesses (Project GOLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 814243; U01PS003304 (NIH); P30MH097488 (NIH)
Record Dates: First submitted 2017-11-01; First posted 2017-11-21 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: HIV; STI; Emotional Disturbances; Mental Disorder
Keywords: Black; Adolescents; Community-based research; Randomized controlled trial; Intervention; Behavioral science
MeSH Terms: conditions — Sexually Transmitted Diseases; Affective Symptoms; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Enrolled participants were randomized to either the targeted intervention group or the attention control group at the diagnostic visit. The permuted-block randomization technique was used with a block size of 4 and a 1:1 allocation ratio. Dr. Alex Hanlon (biostatistics consultant) generated the randomization list using a pseudo-randomizer computer program. The Research Coordinator maintained the spreadsheet for tracking and allocation concealment. To reduce the risk of encountering a floor or ceiling effect with intervention responsiveness, participants were stratified based on their PHQ-9 total scores (none/moderate depression versus moderately severe/severe depression) and gender.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV/STI Prevention Intervention (Experimental): Two-session, small group HIV/STI prevention intervention.
  Interventions: Behavioral: HIV/STI Prevention Intervention
- General Health Control Intervention (Active Comparator): Two-session, small group general health promotion intervention.
  Interventions: Behavioral: General Health Control Intervention

INTERVENTIONS:
Behavioral: HIV/STI Prevention Intervention — The targeted HIV/STI risk reduction intervention was delivered with groups of up to 8 participants through 8, 45-minute modules equally divided over 2 days (4 modules per session). It was designed to enhance participants' knowledge and ability to reduce their risk of HIV/STIs. Grounded in both social/behavioral and cognitive theories, the intervention includes psychoeducation, and was intended to enhance participants' HIV/STI prevention knowledge, attitudes, beliefs and skills in a manner relevant to Black adolescents.
  Arms: HIV/STI Prevention Intervention
Behavioral: General Health Control Intervention — The original Promoting Health among Teens (PHAT) Project was designed to increase knowledge and motivation regarding healthful dietary practices, aerobic exercise, and breast and testicular self-examination, and to discourage cigarette smoking. The 8-hour, 2-session PHAT intervention was shortened to mirror the Project GOLD HIV/STI risk reduction curriculum. This was done to control for the Hawthorne effect and reduce the likelihood that effects of the HIV/STI risk reduction intervention can be attributed to its nonspecific features, including special attention. From an ethical standpoint, adolescents in both conditions received a valuable and engaging health-risk-reduction intervention as opposed to "usual care."
  Arms: General Health Control Intervention

SUMMARY:
Despite advances in HIV/sexually transmitted infection (STI) prevention, Black youth account for the largest number of new HIV infections among heterosexual youth. Having a mental illness contributes to HIV/STI risk among heterosexually active Black youth, as some use sex as a means to manage psychological distress, regulate emotions and receive validation or acceptance. Current intervention models focus on cognitive-behavioral strategies to reduce risk among adolescents; however, these approaches in isolation do not address the psychopathology that further potentiates risk behaviors among adolescents with mental illnesses. This randomized controlled trial evaluated the effects of "Project GOLD", a theoretically-driven, gender and culturally relevant, developmentally and psychologically appropriate HIV/STI risk reduction intervention on the sexual behaviors of Black male and female adolescents in Philadelphia (aged 14-17). In addition to evidence-based HIV/STI preventions strategies (e.g., role playing), Project GOLD includes unique emotion regulation content to address the relationship between psychological distress and HIV/STI risk behaviors.

The research team approached and screened 704 adolescents. Eighty-two participated in the elicitation research activities (e.g., focus groups, intervention dress rehearsal). Another 173 underwent a structured demographic and mental health diagnostic interview to determine RCT eligibility. Project GOLD was then tested with 108 Black youth in comparison to a general health promotion control condition (intervention n = 52; control n = 56). Youth who were not in psychiatric treatment were also included, as the investigators hypothesized that they would also benefit from the targeted psychoeducational content; post-hoc analyses examined differences in the intervention effects based on whether or not youth were in psychiatric treatment. The intervention had high feasibility and acceptability. These findings underscore the need to encourage HIV/STI testing and risk reduction efforts among Black youth, including those with mental illnesses.

DETAILED DESCRIPTION:
This project was approved by the University of Pennsylvania, the Philadelphia Department of Public Health, and the School District of Philadelphia. The primary study site was the University of Pennsylvania. Recruitment took place at public locations in the city of Philadelphia (e.g., recreational centers, community events), Community Behavioral Health (CBH) provider sites, and schools in the School District of Philadelphia.

Phase 1: Team-Building and Elicitation Research (Study aim #1; N = 53). Team building and community engagement were an ongoing process throughout the course of the study. The investigators initially focused on team-building and strengthening ties with collaborators, securing buy-in from key community stakeholders and providers, recruiting 8 members for a youth CAB, and hiring and training project staff. The investigators were committed to the development of an acceptable, practical intervention which could easily be implemented and sustained in the targeted community setting. Therefore, continual feedback from Black adolescents with mental illnesses, CBH providers and research staff was pivotal. Further, Black adolescents in the target demographic and young adults from the community were hired as members of the study team in a capacity building approach to create a pipeline for future HIV/AIDS research investigators and community workers. The investigators also built upon their existent elicitation research with members of the study population. Four mixed gender focus groups were conducted with concurrent open-ended questionnaire administration with Black adolescent males (n= 18) and females (n= 15). The team held meetings with CBH providers and the youth CAB to determine factors associated with HIV/STI risk related sexual behaviors in the population, and the role of psychiatric symptoms, the social determinants of health, gender and culture in sexual risk taking among Black adolescents with mental illnesses. The baseline intervention questionnaire was also piloted with Black adolescent males (n= 10) and females (n= 10) for accuracy; revisions were made based on participant suggestions. Psychometrics of the revised instrument were assessed and results compared to the original version. The qualitative and quantitative data were examined concurrently to explore participants' behavioral, normative and control beliefs, as well as contextual factors, as they relate to HIV/STI risk. Subsequently, this knowledge was used in the design of the targeted intervention.

Phase 2: Intervention Development and Pre-Pilot Testing (Study aim #2; N = 29). The investigators used an iterative process to develop the targeted intervention. They sought feedback from their elicitation participants, youth CAB, and CBH providers at each stage of intervention development. This input was used to ensure accurate interpretation of the study findings, as well as to refine the intervention for relevance and sustainability. The primary outcome of these processes was the development of "Project GOLD", a theoretically-driven, gender and culturally relevant, developmentally and psychologically appropriate behavioral intervention to reduce HIV/STI risk among heterosexually-active Black adolescents receiving outpatient mental health treatment. The intervention name was created by the youth CAB, along with the project logo. The intent in this branding was to foster gender and cultural pride through visually and verbally reinforcing the intervention's tagline: "We are Kings and Queens who make confident and royal decisions". The first pre-pilot testing, or dress rehearsal, of the interventions and all study materials and instruments was conducted with a sample of Black adolescent males (n= 4) and females (n= 4). Participants completed pre- and post-intervention assessments, and the team debriefed with them to solicit their feedback on ways to improve the project. Revisions were made and a new, independent sample of Black adolescent males (n= 3) and females (n= 4) completed the second pre-intervention pilot. The investigators completed the same process for the general health intervention (N = 14). The goals of the intervention pilots were to evaluate whether the interventions were likely to affect the conceptual variables, to evaluate whether the participants viewed the interventions as valuable and engaging, and to ensure the study protocols were relevant to achieve the aims.

Phase 3: Intervention Pilot (Study aims #3 & 4; N = 108). Based on the Phase 2 findings, the final versions of the intervention protocols, materials and instruments were developed and sent for printing. The intervention was piloted with 108 youth; 109 enrolled but one participant was terminated at the baseline visit for eminent suicide risk. Participants were randomized to either Project GOLD (n = 52) or the general health promotion control arm (n = 56). There were five RCT visits: baseline, immediate post, and 3-, 6-, and 12-month follow-up.

RCT Sample, Recruitment and Enrollment. Provider referrals, waiting room encounters, flyers, social media, and teen-focused community events and locations (e.g., talent showcases and game nights; recreational centers) were used to inform potential participants about the study. As part of the investigators' community engagement mission, the research team hosted programs and/or partnered with local community-based organizations to promote HIV/STI awareness and encourage testing among youth. In an effort to increase study enrollment, staff members also screened interested youth for eligibility at these events. The programs took place in reserved campus space at the University of Pennsylvania, or a public community space as approved (e.g., local YMCA or recreation center). Eligibility was determined using a structured screening script either in person or by telephone. All study visits took place at one of the sites where participants were recruited, at the University of Pennsylvania in a private conference room, or in a private conference room at a community-based organization near where participants are recruited (e.g., recreation center). No data collection occurred at any School District schools or property as a condition of their IRB approval. For the RCT, participants registered with the study coordinator, were assessed by a research team member using an electronic version of the Patient Health Questionnaire-9 (PHQ-9), provided a urine specimen, had their mouths swabbed for the rapid HIV test, and completed the self-administered sexual risk behavior questionnaire in a private, quiet room.

Assent versus Consent. In the state of Pennsylvania, adolescents between the ages of 14 to 17 can autonomously make decisions about their sexual and mental health assessment and treatment. "…[I]f a minor is able to consent to medical, dental and health services under state law, the minor is also able to consent to take part in medical research" (pg. 9). Therefore, youth aged 14 to 17 provided consent to participate in the research without parental permission. Initial disagreements among the approving IRBs, however, lead to substantial protocol delays. The investigators agreed to exclude (or withdraw from participation) any adolescent whose parent/guardian is aware of/finds out about the study and indicates that they do not want their son or daughter to participate in the research. This was honored if a participant shared that his or her parent/guardian expressed to them that they did not want them in the study, or if the parent/guardian directly contacted a member of the research team to state they did not want their son or daughter to be involved.

Procedures for Consent/Assent & Diagnostic Assessment. Adolescents who were preliminarily eligible were scheduled for their first study visit to undergo a 30-minute diagnostic assessment using the MINI to ascertain psychiatric diagnosis and rule out exclusionary disorders. Trained study personnel conducted all of the diagnostic assessments. Based on the diagnostic assessment, adolescents were excluded if they: 1) had a psychotic disorder, or disorder with psychosis, 2) were cognitively impaired, or 3) their current treatment required hospitalization. Eligible participants immediately participated in a brief, 10-minute structured demographic interview. The interview was used to obtain locator information to follow participants over the course of the study, as well as to elicit information regarding referral source, demographics, and clinical data (i.e. psychiatric and medical history). The structured diagnostic and demographic interviews took approximately 40 minutes. At the end of the structured interviews, participants were scheduled for their second study visit which included the baseline assessment and first intervention session.

Procedures for Enrollment, Randomization & Intervention Trial. At the second study visit, participants completed the electronic baseline assessments (Intervention Baseline Questionnaire which includes the Background Information Questionnaire and PHQ-9) and provided urine specimens for STI testing. When the urine specimens were obtained, all participants signed a medical release form so that the study's Nurse Practitioner could receive the STI test results and confirm treatment for positive results with the health centers or chosen providers. They then immediately attended the first intervention session following these procedures. Randomization to either the targeted intervention or treatment control group occurred at the diagnostic visit. Where feasible, intervention and control group sessions ran concurrently at the same site; if the sessions could not be run on the same day, intervention and control group sessions were delivered within the same week at each site, or as close as possible thereafter. Participants attended the second intervention session (their third study visit) two weeks after the first intervention session. Immediately following the second/final intervention session they completed post-intervention measures, had their mouths swabbed for a rapid HIV test, and received their HIV/STI results. In accordance with the CDC's Revised Recommendations for HIV Testing of Adults, Adolescents, and Pregnant Women in Health Care Settings, HIV screening was provided for all participants unless a participant expressly refused to take an HIV test (59.3% consented to HIV testing). Thus, study participants were offered HIV testing but not required to consent to testing to participate in the study. Participants also returned for post-intervention follow-up visits 3-, 6-, and 12-months after the date of their final intervention session. At each study visit, participants registered with the study coordinator, were screened with the electronic PHQ-9 and had all appropriate labs collected. They were then seated in a quiet room and provided with the electronic, self-administered Background Information Questionnaire.

No adolescents tested positive for HIV over the course of the study. Those who tested positive for another STI were permitted to stay in the study. The study Nurse Practitioner notified participants of their baseline STI results at the end of the final intervention session, and participants received subsequent notifications by phone within 2-weeks after each of the 3 follow-up time points. Individuals who tested positive for an STI were referred to receive free treatment through the Philadelphia Health Department at the designated STI control health centers (Health Centers #1 [500 S. Broad St.] and #5 [1900 N. 20th St.]). Individuals who tested positive for an STI and fail to be located, did not comply with returning to the study site, or who failed to seek clinical treatment through an alternative provider, were reported to the City of Philadelphia Department of Public Health, as required by the City of Philadelphia.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 17 years old
* Self-identify as Black (inclusive of African American, Caribbean-American, etc.)
* Have ever had vaginal sex
* Able to speak, read and write in the English language
* Able to provide signed informed consent/assent
* Plan to be in the Philadelphia area for the next 12 months.

Exclusion Criteria:

* Diagnosis of a psychotic disorder (i.e. Schizophrenia) or a disorder with psychotic features (ascertained by the MINI)
* Cognitive deficit that would impair ability to complete study procedures
* Actively suicidal (ascertained through the Columbia-Suicide Severity Rating Scale [C-SSRS]) or requiring hospitalization
* Unstable contact information (i.e. homeless or no permanent address, or no land line or mobile phone)

Participants were not excluded for concurrent use of herbal remedies, mineral supplements, or psychopharmacologic therapies, however these factors will be controlled for in the data analyses.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline consistent condom use at 12 months | 12 months
  This dichotomous variable was defined by the comparison of the number of protected intercourse acts and the number of intercourse acts. Participants who report at least one intercourse act and whose number of reported protected acts equals their number of acts use condoms during 100% of intercourse acts and will be defined as practicing consistent condom use. Participants who report at least one intercourse act and whose reported number of protected acts is less than their number of acts will be coded as not practicing consistent condom use.

SECONDARY OUTCOMES:
Change from baseline number of sexual partners at 12 months | 12 months
  A continuous variable was calculated in response to questions about the number of sexual partners participants had in the past 12-months.
Change from baseline laboratory confirmed STIs at 12 months | 12 months
  Diagnosis of Chlamydia trachomatis (CT) and Neisseria gonorrhea (GC) was made based on DNA amplification tests on urine specimens at baseline and follow-up. Participants provided an on-site first-void urine specimen of approximately 15 to 20 cc. Dichotomized as positive STI result yes/no.
Change from baseline HIV Diagnosis at 12 months | 12 months
  Diagnosis of HIV was made based by laboratory confirmation following a positive OraQuick Advance Rapid HIV-1/2 antibody test at baseline and follow-up. This rapid HIV antibody tests detects antibodies to HIV-1 and HIV-2 within 20 minutes (Oraquick; Orasure Technologies, Inc.). Saliva was swabbed between the teeth and upper and lower gum by a certified HIV tester and counselor from the partner ASO. Dichotomized as HIV positive yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette M Brawner, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
For other investigators interested in using the data for secondary data analysis purposes (e.g., students, faculty), we will develop a data use agreement with specific guidelines associated with the parent study. This will include information related to confidentiality of the data and human subjects' protection, as well as the acknowledgement of our study in all publications and presentations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available starting 6 months after publication of the main study outcomes, and remain available.
Access Criteria: Dr. Brawner will be responsible for making de-identified data collected from the study available to other investigators upon their request. Interested investigators will be able to request formal access to the data from Dr. Brawner in writing, and the request will be reviewed within a timely manner and data will be provided.

REFERENCES:
- [Background] Brawner BM, Jemmott LS, Wingood G, Reason J, Mack N. HIV/STI Prevention Among Heterosexually Active Black Adolescents With Mental Illnesses: Focus Group Findings for Intervention Development. J Assoc Nurses AIDS Care. 2018 Jan-Feb;29(1):30-44. doi: 10.1016/j.jana.2017.09.008. Epub 2017 Sep 28. PMID 29037602